CLINICAL TRIAL: NCT00558129
Title: Prospective Randomized Trial Comparing X-STOP® Interspinous Process Decompression® System Versus Laminectomy for Treatment of Neurogenic Intermittent Claudication
Brief Title: Effects of X-STOP® Versus Laminectomy Study
Acronym: EXELS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Spine LLC (Industry)
Responsible Party: Sponsor
Organization: Medtronic Spinal and Biologics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LSS0702
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2012-01

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar Spinal Stenosis; X-STOP® IPD; Interspinous process decompression; Neurogenic Intermittent Claudication
MeSH Terms: conditions — Spinal Stenosis | interventions — Laminectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational (Experimental): X-STOP® PEEK IPD
  Interventions: Device: X-STOP®
- Control (Active Comparator): Laminectomy
  Interventions: Procedure: Laminectomy

INTERVENTIONS:
Device: X-STOP® — Surgical implantation of X-STOP IPD device
  Other Names: X-STOP® PEEK IPD
  Arms: Investigational
Procedure: Laminectomy — Standard laminectomy techniques will be used and may include laminotomy, foraminotomy and/or laminectomy as appropriate. In some cases at the discretion of the treating physician, fusion may indicated to stabilize the segment.
  Arms: Control

SUMMARY:
To determine if the effectiveness of the X-STOP® implant is equivalent (non-inferior) to that of conventional laminectomy in patients with lumbar spinal stenosis as measured by the Zurich Claudication Questionnaire.

DETAILED DESCRIPTION:
The clinical study described herein aims to compare surgical outcomes of X-STOP® Interspinous Process Decompression® (IPD) system implantation and conventional laminectomy in subjects requiring surgical intervention due to symptoms of lumbar spinal stenosis (LSS) and a confirmed diagnosis on MRI, X-ray or CT. Patients with LSS meeting entry criteria will be randomized to either X-STOP® IPD or laminectomy treatment. Patients will remain blinded to the procedure received. The primary study outcome is group differences in the Zurich Claudication Questionnaire (ZCQ) at 12 months post-operative. In addition, each subject will undergo follow-up assessment at 2 weeks and 2, 12 and 24 months post-operative. The secondary objective is to compare safety profiles and the radiographic outcomes between groups using pre- and post-operative MRI and flexion/extension X-rays, to measure changes in canal and neuroforaminal cross sectional areas and spinal stability, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 50
2. Has completed at least 6 months of conservative therapy which may include but is not limited to epidural steroid injection, oral steroids, NSAIDS, analgesics, physical therapy, and/or spinal manipulation.
3. Symptoms of leg/buttock/groin pain with or without back pain that are exacerbated by lumbar extension and relieved in flexion. If back pain is also present it must be partially relieved when the patient flexes.
4. Diagnosis of NIC due to lumbar stenosis at 1 or 2 lumbar levels confirmed by X-ray, MRI or CT.
5. Subject is a surgical candidate with disease severity justifying that BOTH laminectomy and X-STOP IPD placement are clinically appropriate treatment options.
6. Baseline score of >2.0 in the Physical Function domain of the Zurich Claudication Questionnaire (ZCQ). Because this is a post-market study, the Inclusion Criteria are consistent with FDA approved X-STOP indication for use (moderately impaired physical function), which requires a ZCQ physical function score of >2.0.
7. Subject is able to walk at least 50 feet.
8. Subject is willing and able to comply with required follow-up testing and expected to be physically able to return for evaluation at scheduled follow-up visits.
9. Subject is able to understand the risks and benefits of participating in the study.
10. Subject understands and has signed the study informed consent form.

Exclusion Criteria:

1. Spinal stenosis involving more than 2 lumbar levels.
2. Any previous lumbar spine surgery.
3. Subject has unremitting pain in any spinal position or axial back pain only without leg/buttock/groin pain.
4. Evidence that subject's symptoms are due to vascular claudication.
5. Subject has significant instability of the lumbar spine, e.g., isthmic spondylolisthesis or degenerative spondylolisthesis greater than Grade 1 (on a scale of 1 to 4).
6. Subject has an ankylosed segment at the affected level(s).
7. Subject has significant scoliosis (Cobb angle is greater than 25 degrees).
8. Subject has cauda equina syndrome defined as neural compression causing neurogenic bowel (rectal incontinence) or bladder (bladder retention or incontinence) dysfunction.
9. Subject has a fixed motor deficit or known peripheral neuropathy.
10. Subject has a degenerative neurologic disease.
11. Subject has any mass lesions (e.g. disc herniations, synovial cysts, spinal tumors).
12. Any evidence of spinal or systemic infection.
13. Subject has a history of spinous process fracture or pars interarticularis fracture.
14. Subject has history or radiographic evidence of 1 or more osteoporotic fractures (e.g., vertebral, hip, wrist) OR subject has severe osteoporosis of the spine or hip, defined as bone mineral density (BMD) in the spine or hip more than 2.5 SD below the mean of adult normals. If the Investigator suspects osteoporosis, a DEXA scan should be done.
15. Subject has a known allergy to the implant materials (this includes titanium or titanium alloy and polyetheretherketone for X-STOP IPD).
16. Subject has a bleeding disorder or an active systemic disease such as HIV, hepatitis, etc.
17. Subject has any medical condition that would limit availability for follow-up.
18. Subject has a recent history of narcotic abuse (i.e., within last 3 years).
19. Subject is immunologically suppressed, or has received or is receiving 7.5 milligrams prednisone (or equivalent) daily for more than six months immediately prior to enrollment.
20. Subject is currently involved in a study of another investigational product that may affect the outcome of this study.
21. Subject is not able to undergo MRI or tolerate closed MRI scanning. Subject is pregnant or of child-bearing potential and not currently on adequate birth control method.
22. Subject is pregnant or of child-bearing potential and not currently on adequate birth control method.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Zurich Claudication Questionnaire (ZCQ) | 1 year post-operative

SECONDARY OUTCOMES:
ZCQ symptom severity, physical function and satisfaction; pain rating; quality of life (SF-36®); operative data; canal, subarticular and neuroforaminal measurements on MRI; spinal stability using flexion/extension (serious adverse events) | Out to 2 years postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Volker Sonntag, MD, Principal Investigator — Barrow Neurological Institute, St. Joseph's Hospital and Medical Center